CLINICAL TRIAL: NCT07042763
Title: Subciliary Closure in Orbital Fracture: Comparison Between Cutaneous and Cutaneous-periosteal Suture
Brief Title: Subciliary Closure in Orbital Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, Principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-1301-112.
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Orbital Floor Fractures; Surgical Wound Closure Techniques; Subciliary Surgical Approach; Postoperative Complications in Maxillofacial Surgery
Keywords: Orbital Fractures; Eyelid Diseases; Surgical Wound Dehiscence; Suture Techniques; Postoperative Complications
MeSH Terms: conditions — Orbital Fractures; Eyelid Diseases; Surgical Wound Dehiscence; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, randomized, prospective surgical trial. Patients were assigned to one of two different closure techniques during orbital floor fracture repair.
Masking Description: Not applicable. The surgical technique was visible to both care providers and patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cutaneous Suture (Active Comparator): Subciliary incision closed with 5-0 nylon skin sutures only. No periosteal sutures were used.
  Interventions: Procedure: Cutaneous Suture
- Periosteal Suture (Experimental): Subciliary incision closed with both periosteal (4-0 Vicryl) and cutaneous (5-0 nylon) sutures.
  Interventions: Procedure: Cutaneous Suture; Procedure: Periosteal Suture

INTERVENTIONS:
Procedure: Cutaneous Suture — Subciliary incision followed by closure using skin sutures only. The skin was closed with 5-0 nylon using subdermal interrupted sutures. No closure of the periosteal plane was performed.
Procedure: Periosteal Suture — Subciliary incision followed by closure of both the periosteum and skin layers. The periosteum was closed with absorbable 4-0 Vicryl sutures, and the skin was closed with 5-0 nylon using subdermal sutures.
  Arms: Periosteal Suture

SUMMARY:
Title: Subciliary Closure in Orbital Fractures: A Comparison Between Cutaneous and Cutaneo-Periosteal Sutures

Brief Summary:

This prospective, experimental, and comparative study evaluated the impact of two different subciliary wound closure techniques in patients undergoing surgical repair of orbital floor fractures. The study was conducted at a tertiary care center in Mexico from July to October 2024 and included 100 adult patients with isolated orbital floor fractures, excluding LeFort-type fractures.

Participants were randomized into two groups: Group 1 received skin-only subciliary sutures, while Group 2 underwent closure using both cutaneous and periosteal sutures. The objective was to determine whether the addition of periosteal sutures influenced the rate of common postoperative complications, including eyelid retraction, ectropion, and the need for surgical reintervention.

Postoperative evaluations were conducted on days 8, 15, and 30. Outcomes measured included incidence of eyelid retraction, ectropion, reoperation rate, and any association with comorbidities such as smoking, diabetes, hypertension, or substance use.

The study found a statistically higher incidence of eyelid retraction in the group with combined periosteal and cutaneous closure at postoperative day 8 (16% vs. 2%, p=0.014) and day 15 (20% vs. 6%, p=0.037). However, no significant differences were noted in rates of ectropion or reintervention. Smoking, the most common comorbidity in the cohort, was not associated with a higher rate of complications.

This study suggests that skin-only closure may be preferable in subciliary orbital approaches, as it is associated with fewer cases of eyelid retraction without increasing the risk of other complications.

DETAILED DESCRIPTION:
Orbital floor fractures are among the most frequent midfacial injuries and are typically managed through surgical reconstruction via a subciliary or transconjunctival approach. Despite the frequency of these procedures, there is limited evidence evaluating the role of closure technique-specifically, whether adding periosteal sutures to cutaneous closure affects postoperative outcomes.

This study was designed to investigate whether dual-layer closure (periosteum and skin) influences the incidence of lower eyelid complications such as retraction, ectropion, and need for reoperation, compared to skin-only closure in patients treated via the subciliary approach.

Eligible participants were adults diagnosed with orbital floor fractures indicated for open surgical reduction and internal fixation. All procedures were performed by experienced surgical teams following a standardized protocol. Patients were followed for one month after surgery, and clinical outcomes were systematically assessed at three timepoints (days 8, 15, and 30 postoperatively).

The primary outcome was the presence or absence of eyelid retraction. Secondary outcomes included incidence of ectropion, need for surgical revision, and association of complications with risk factors such as smoking, diabetes, and hypertension.

This trial addresses a clinical gap by evaluating the impact of periosteal suturing in orbital trauma surgery. Findings may help guide surgeons in optimizing closure techniques to improve functional and aesthetic outcomes while minimizing postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Diagnosis of orbital floor fracture requiring surgical intervention
* Treatment planned through subciliary surgical approach
* Ability to attend scheduled follow-up visits at postoperative day 8, 15, and 30
* Signed informed consent obtained prior to study inclusion

Exclusion Criteria:

* Fractures involving Le Fort I, II, or III patterns
* History of prior orbital surgery or trauma on the affected side
* Presence of active ocular infection or orbital cellulitis
* Uncontrolled systemic disease (e.g., decompensated diabetes, bleeding disorders)
* Pregnant or breastfeeding women
* Known non-compliance with postoperative care or follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Lower Eyelid Retraction | Postoperative Day 8, Day 15, and Day 30
  The presence of clinically observable lower eyelid retraction following subciliary surgical closure will be evaluated through physical examination. Eyelid retraction is defined as the inferior displacement of the lower eyelid margin exposing the sclera.

SECONDARY OUTCOMES:
Incidence of Ectropion | Postoperative Day 8, Day 15, and Day 30
  Ectropion will be assessed by clinical inspection, defined as outward turning of the eyelid margin resulting in loss of eyelid-globe contact.
Need for Surgical Reintervention | Within 30 days of initial surgery
  Participants requiring a second surgical procedure due to complications associated with eyelid retraction, ectropion, infection, or other closure-related issues will be recorded.

OTHER OUTCOMES:
Correlation Between Smoking Status and Eyelid Retraction | From enrollment to postoperative day 30
  This outcome assesses whether active smoking is associated with an increased incidence of lower eyelid retraction following subciliary surgical closure. Eyelid retraction will be evaluated by physical examination and defined as the inferior displacement of the eyelid margin exposing the sclera.
Correlation Between Smoking Status and Ectropion | From enrollment to postoperative day 30
  This outcome evaluates whether active smoking correlates with the incidence of ectropion after orbital fracture repair. Ectropion is defined as outward turning of the eyelid margin with loss of eyelid-globe contact, assessed by clinical inspection.
Correlation Between Smoking Status and Need for Surgical Reintervention | From enrollment to 30 days after initial surgery
  This outcome assesses whether active smoking increases the need for a secondary surgical procedure due to complications such as eyelid retraction, ectropion, or wound-related problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Especialidades del Centro Médico Nacional de Occidente (CMNO) - IMSS, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data due to institutional restrictions and the non-pharmacologic nature of the intervention.

REFERENCES:
- [Background] Cornelius CP, Mayer P, Ehrenfeld M, Metzger MC. The orbits--anatomical features in view of innovative surgical methods. Facial Plast Surg. 2014 Oct;30(5):487-508. doi: 10.1055/s-0034-1394303. Epub 2014 Nov 14. PMID 25397705
- [Background] Committeri U, Arena A, Carraturo E, Austoni M, Germano C, Salzano G, De Riu G, Giovacchini F, Maglitto F, Abbate V, Bonavolonta P, Califano L, Piombino P. Incidence of Orbital Side Effects in Zygomaticomaxillary Complex and Isolated Orbital Walls Fractures: A Retrospective Study in South Italy and a Brief Review of the Literature. J Clin Med. 2023 Jan 20;12(3):845. doi: 10.3390/jcm12030845. PMID 36769492
- [Background] Turvey TA, Golden BA. Orbital anatomy for the surgeon. Oral Maxillofac Surg Clin North Am. 2012 Nov;24(4):525-36. doi: 10.1016/j.coms.2012.08.003. PMID 23107426